CLINICAL TRIAL: NCT06424340
Title: A Phase I/II Trial of MB-dNPM1-TCR.1 in HLA-A*02:01-positive Patients With Relapsed or Refractory NPM1-mutated AML to Determine Safety and Obtain First Data on Efficacy
Brief Title: MB-dNPM1-TCR.1 in Relapsed/Refractory AML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2020-358
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MB-dNPM1-TCR.1 (Experimental): Biological: MB-dNPM1-TCR.1
  Interventions: Biological: MB-dNPM1-TCR.1

INTERVENTIONS:
Biological: MB-dNPM1-TCR.1 — T Cell Receptor (TCR) T cell therapy

SUMMARY:
The goal of this Phase I/II, single arm, prospective, open label, dose escalation trial is to assess safety, feasibility and efficacy of ex vivo expanded autologous T cells genetically modified to express a T cell receptor (TCR) specific for dNPM1 peptides restricted to human leukocyte antigen (HLA) A*02:01 in patients with relapsed or refractory AML.

DETAILED DESCRIPTION:
The investigational medicinal product (IMP) MB-dNPM1-TCR.1 is designed to effectively target malignant myeloid cells in patients suffering from relapsed or refractory Acute Myeloid Leukemia (AML) with mutated Nucleophosmin. Autologous T cells will be genetically engineered using a lentiviral vector to express a T cell receptor (TCR) specific for certain dNPM1 peptides restricted to human leukocyte antigen (HLA) A*02:01. The dNPM1-TCR transduced T cells target specifically the HLA/dNPM1 peptide complex on the cell surface of leukemic myeloid cells and eliminate these. During the treatment, the patients will undergo a leukapheresis, a lymphodepleting chemotherapy and an administration of the expanded dNPM1-TCR transduced T cells.

Phase I: Since this is a first in human trial the primary goal in phase I is to establish the recommended dose of MB-dNPM1-TCR.1 for phase II. We assess the maximum tolerated dose (MTD) with toxicity defined as patients experiencing dose limiting toxicity (DLT) until day 28 after infusion of MB-dNPM1-TCR.1. Therefore a BOIN trial design will be used to guide dose escalation and de-escalation decisions in phase I.

Phase II: The second phase will evaluate the efficacy and safety in patients treated with the recommended dose from phase I. The phase II part follows a Simon's 'minimax' two stage design.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients must be able to understand and be willing to give signed informed consent
3. Relapsed or refractory acute myeloid leukemia (last disease staging within 4 weeks prior to screening) without standard treatment options defined as:

   * No morphological CR after at least two courses of intensive chemotherapy, decitabine or other standard therapy or
   * MRD positive after at least two courses of intensive chemotherapy and not eligible for allogeneic stem cell transplantation or
   * Relapsed bone marrow or blood disease after CR after first line treatment and not eligible to undergo allogeneic stem cell transplantation or
   * Bone marrow or blood relapse, non-response or MRD positivity after allogeneic stem cell transplantation and not eligible to receive Donor Lymphocyte Infusion (DLI) according to local standards, relapse after DLI.
4. Positive for HLA-A*02:01 according to genotyping results.
5. AML has NPM1 mutation which is recognized by dNPM1-TCR.1 and for which a specific Q-PCR is available for disease monitoring.
6. Number of circulating WBC above 1x109/L with less than 20% leukemic blasts and at least 0.3x109 T cells/L and 0.03 x 109 CD8+ T cells/L.
7. Life expectancy of at least 3 months.
8. ECOG performance status 0-3.
9. Negative pregnancy test in women of childbearing potential.
10. For fertile men and women, agreement to use highly effective contraceptive methods during the trial.

Exclusion Criteria:

1. Pregnant or breast feeding women.
2. Active infection with HIV-1, HIV-2, HBV, HCV, HTLV-I, HTLV-II, SARS-CoV-2 or Treponema Pallidum.
3. Any clinically significant, advanced or unstable disease or inadequate main organ function that may put the patient at increased risk for severe complications of trial participation at the discretion of the investigator.
4. Use of systemic immune suppression including, but not limited to:

   immunosuppressive agents such as cyclosporine or corticosteroids (at an equivalent dose of 0.5 mg prednisone/kg body weight per day, or higher). Inhaled steroid and physiological replacement for adrenal insufficiency are allowed.
5. Unwillingness or inability to comply with procedures required in this clinical trial protocol.
6. Uncontrolled central nervous system (CNS) disease.
7. Uncontrolled life-threatening infections or uncontrolled disseminated intravascular coagulation; however, if these problems resolve, the start of treatment can be initiated on a delayed schedule.
8. Subjects currently on any other IMP (including within the last 30 days before start of treatment).
9. Current use of high dose immunosuppression for immune disorders interfering with T cell function (on discretion of the investigator).
10. Known hypersensitivity against any drug of the mandatory trial procedures.
11. Serum creatinine ≥ 2.0 × ULN or eGFR < 30 mL/min calculated according to the modified MDRD formula.
12. BMI ≥40
13. Has received vaccination with live vaccines 6 weeks prior to treatment
14. Major surgery less than 30 days before start of treatment.
15. Committal to an institution on judicial or official order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint Phase I | day 28
  Maximum tolerated dose (MTD), as identified by a Bayesian Optimal Interval (BOIN) design at a target toxicity rate of 30%, with toxicity defined as patients experiencing dose limiting toxicity (DLT) until day 28 (week 4) after infusion of MB-dNPM1-TCR.1.
Primary endpoint Phase II | week 12
  BOR rate to the treatment with MB-dNPM1-TCR.1 assessed at any time within the first 3 months (12 weeks) after infusion as described above.

SECONDARY OUTCOMES:
Persistence | from day 6 to week 96
  Percentage and total number of MB-dNPM1-TCR+ cells in peripheral blood and/or bone marrow over time.
Best objective response (BOR) | week 12
  Best objective response (BOR) during 12 weeks after infusion of MB-dNPM1-TCR.1. BOR is defined in relation to disease activity before thawing the leukapheresis for manufacturing (day -18 and -15).
Overall survival (OS) | up to week 96
  Overall survival (OS) defined as the time between the date of infusion of MB-dNPM1-TCR.1 and the date of death from any cause.
Progression-free survival (PFS) | up to week 96
  Progression-free survival (PFS) defined as the time between the date of infusion of MB-dNPM1-TCR.1 and the date of objective disease progression or death from any cause whichever occurs first.
Duration of response (DOR) | up to week 96
  Duration of response (DOR), defined as the time between the date of the first objective response (CRMRD- CR, CRi, MLFS, PR, SD) and the date of assessment of relapse or the date of death due to AML, whichever occurs first.
Safety and toxicity | up to week 96
  Safety and toxicity assessment of MB-dNPM1-TCR.1 per (serious) adverse events ((S)AE) reporting.
Feasibility to manufacture | Day 0
  Proportion of thawed apheresis products, from which MB-dNPM1-TCR.1 drug products are produced.

CONTACTS AND LOCATIONS:
Overall Officials: C.J.M. Halkes, Dr, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No